CLINICAL TRIAL: NCT04513587
Title: CBT-Based Weight Loss Treatment Model in Obese Patients With Comorbid Depression. Effect on Eating Behavior, Weight Loss, Mood, and Risk of Coronary Artery Disease and Diabetes.
Brief Title: The Effect and Applicability of CBT-Based Weight Loss Treatment Model in Obese Patients With Comorbid Depression in Health Care
Acronym: PsyCognObe2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Collaborators: University of Oulu (Other); Jyväskylä Central Hospital (Other); Oulu University Hospital (Other); University of Eastern Finland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 510RA21
Record Dates: First submitted 2019-08-28; First posted 2020-08-14 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Obesity; Depression; Cognitive Behavioral Therapy; Weight Loss
MeSH Terms: conditions — Obesity; Depression; Weight Loss

STUDY DESIGN:
Intervention Model Description: Randomized intervention study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT-Based Weight Loss Model (Experimental): CBT- Based weight loss model
  Interventions: Behavioral: CBT-based weight loss model
- Control (Active Comparator): Usual Care
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: CBT-based weight loss model — Methods of cognitive behavioral psychotherapy
  Arms: CBT-Based Weight Loss Model
Behavioral: Control — Treatment as usual
  Arms: Control

SUMMARY:
The aim of this study is find out how CBT-based weight loss program affects on eating behavior, weight loss, mood symptoms and risk for coronary heart diseases and type 2 diabetes and applicability of the program to obesity treatment among patients with comorbid depression. Our hypothesis is that the CBT-based intervention improves long-term weight management results and supports positively the change in eating behavior and the risk for CHD on type 2 DM.

The study is randomized controlled one-year intervention study with 1 year follow-up. Study subjects are adult obese (BMI>35) subjects with comorbid depression. Number of randomized study subjects will be 80, 40 in intervention group, 40 in control group.

Intervention group will proceed through a 52-week CBT-based weight loss group intervention. The aim of the intervention is to modify eating behavior and lifestyle factors affecting weight and weight maintenance. There will be 22 group counselling of 90 minutes divided in five modules and also three individual person-centered counselling visit, during which participants had an opportunity to discuss their personal concerns about diet and weight loss plan. Control group will receive the usual care of obesity in Kuopio University hospital. (4-8 individual 45-minute visit conducted by dieticians)

Study visits are at baseline and one and 2 years after baseline. For example eating behavior, health behavior, motivation and depression are studied with questionnaires. Weight, waist circumference, height and blood pressure are measured. Laboratory tests (lipid, glucose etc) are taken.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Diagnosed depression ( F32.0, F32.1, F32.2, F33.0, F33.1, F33.2)
* BMI > 35

Exclusion Criteria:

* Psychotic disorder, schizoaffective disorder, psychotic depression or bipolar disorder
* Severe current substance abuse
* Serious psychiatric condition (i.e self-destructive or impulsive behavior)
* Clinically significant illness contraindicating weight loss (i.e cancer or severe heart disease)
* Simultaneous participation in another weight loss program
* Severe vision, hearing, motoric deficiency

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 80 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Weight | baseline and change from baseline to 1 year and 2 years
  Measured by scale on baseline, 1 year and 2 years
Change in Lipids | baseline and change from baseline to 1 year and 2 years
  Measured by laboratory analyses (total cholesterol,High-density lipoprotein, Low-density lipoprotein, Triglyserides
Change in Blood glucose | baseline and change from baseline to 1 year and 2 years
  Measured by laboratory analyses
Change in c-reactive protein level | baseline and change from baseline to 1 year and 2 years
  Measured by laboratory analyses
Change in Glycated hemoglobin (HbA1c) | baseline and change from baseline to 1 year and 2 years
  Measured by laboratory analyses
Change in Waist circumference | baseline and change from baseline to 1 year and 2 years
  Measured by tape measure on baseline, 1 year and 2 years

SECONDARY OUTCOMES:
Change in Eating behavior assessed by TFEQ-18 questionnaire | baseline and change from baseline to 1 year and 2 years
  Three Factor Eating questionnaire-18 measures three eating behavior traits: emotional eating, cognitive restraint and uncontrolled eating.
Change in Eating behavior assessed by BES-questionnaire | baseline and change from baseline to 1 year and 2 years
  BES -questionnaire assess binge eating symptoms.
Change in Intuitive Eating behavior | baseline and change from baseline to 1 year and 2 years
  assessed by IES2 (Intuitive Eating Scale) questionnaire,
Change in Physical acitivity | baseline and change from baseline to 1 year and 2 years
  assessed by questionnaire assessing physical activity
Change in Sleep | baseline and change from baseline to 1 year and 2 years
  assessed by questionnaire
Change in Use of alcohol and tobacco | baseline and change from baseline to 1 year and 2 years
  assessed by questionnaire
Previous weight loss | baseline
  assessed by questioinnaire
Change in Mood | baseline and change from baseline to 1 year and 2 years
  assessed by BDI (Beck Depression Inventory) questionnaire
Change in Anxiety | baseline and change from baseline to 1 year and 2 years
  assessed by BAI (Beck Anxiety Inventory) questionnaire
Change in Quality of life | baseline and change from baseline to 1 year and 2 years
  Assesed by 15D questionnaire
Change in Self-efficacy: questionnaire | baseline and change from baseline to 1 year and 2 years
  assessed by WEL questionnaire
Change in Sense of coherence | baseline and change from baseline to 1 year and 2 years
  assesed by SOC13 (Sense of Coherence) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Anna-Maria Teeriniemi, PhD, Principal Investigator — Kuopio University Hospital
Locations (1):
- Kuopio University Hospital, Kuopio, Finland

IPD SHARING:
Plan to Share IPD: No